CLINICAL TRIAL: NCT00002263
Title: A Pilot Study to Evaluate the Effects of Subcutaneously Administered Recombinant Human Granulocyte-Macrophage Colony Stimulating Factor in Pediatric HIV-Infected Patients With Neutropenia Secondary to Azidothymidine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sandoz (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 067B; 206
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-01

CONDITIONS: HIV Infections; Cytopenias
Keywords: Pilot Projects; Neutropenia; Granulocyte-Macrophage Colony-Stimulating Factor; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — HIV Infections; Cytopenia; Neutropenia; Acquired Immunodeficiency Syndrome | interventions — Zidovudine; sargramostim

INTERVENTIONS:
Drug: Zidovudine
Drug: Sargramostim

SUMMARY:
To assess the safety and efficacy of subcutaneous sargramostim ( granulocyte-macrophage colony-stimulating factor; GM-CSF ) in increasing and maintaining the granulocyte count in HIV-infected children who have developed granulocytopenia as a result of continuous intravenous ( CIV ) zidovudine ( AZT ). To assess the short-term and long-term effects of concomitant GM-CSF on other hematologic parameters. To assess the potential therapeutic benefit of concomitant GM-CSF and AZT on the natural history of HIV infection and associated infectious complications.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine (AZT) on NIAID 86-C-175.

Patients must have:

* Diagnosis of perinatal or transfusion acquired AIDS or AIDS related complex.
* Granulocytopenia (< or = to 800 cells/mm3) associated with the administration of AZT on protocol NIAID 86-C-175.
* Life expectancy > 3 months.
* Functioning indwelling central venous access device in place.

Prior Medication:

Allowed within 48 hours of study entry:

* Prophylactic antibiotics.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Critically ill or clinically unstable.
* Significant, active opportunistic or other infection requiring specific drug therapy at time of study entry.
* Ongoing IV alimentation.
* Uncorrected nutritional deficiencies that may contribute to anemia and/or leukopenia.
* Past history of or current evidence for any chronic hematologic disorder other than hemophilia A or B, anemia of chronic disease or anemia related to HIV infection.
* Malignancy likely to require systemic treatment during study.

Patients with the following are excluded:

* Critically ill, clinically unstable, or with concomitant diseases listed in Patient Exclusion Co-existing Conditions.
* Hypersensitivity to zidovudine (AZT) or any other nucleoside analog.

Prior Medication:

Excluded within 48 hours of study entry:

* Antibiotics.
* Excluded within 30 days of study entry:
* Antiretroviral agents other than zidovudine (AZT).
* Acyclovir.
* Ganciclovir.
* Any investigational drug.
* Immunomodulating drugs.
* Cytolytic chemotherapeutic agents.
* Corticosteroids.
* Immunoglobulin preparations.
* Excluded within 4 months of study entry:
* Suramin.

Prior Treatment:

Excluded within 6 months of study entry:

* Bone marrow transplantation.
* Excluded within 4 weeks of study entry:
* Lymphocyte transfusions.
* Radiation therapy.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child

CONTACTS AND LOCATIONS:
Locations (1):
- Natl Cancer Institute / HIV / AIDS Malignancy Branch, Bethesda, Maryland, United States